CLINICAL TRIAL: NCT05133180
Title: A 4-week, Phase III, Multicenter, Double-masked, Vehicle-controlled Clinical Study to Evaluate Safety and Efficacy of Oxervate® (Cenegermin) 20 mcg/mL Ophthalmic Solution vs Vehicle in Severe Sjogren's Dry Eye Disease
Brief Title: Safety and Efficacy Study on Cenegermin (Oxervate®) vs Vehicle in Severe Sjogren's Dry Eye Disease (PROTEGO-1 Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NGF0121; 2021-003346-21 (EudraCT Number)
Record Dates: First submitted 2021-11-15; First posted 2021-11-24 (Actual); Results first posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-05

CONDITIONS: Dry Eye
Keywords: Sjorgen's dry eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — cenegermin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: double-masked study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oxervate (Experimental): One drop of cenegermin 20 mcg/mL (rhNGF 20 mcg/mL) in the pharmaceutical form of ophthalmic sterile solution was instilled in both eyes three times daily (TID), every six hours.
  Interventions: Drug: Oxervate
- Vehicle (Placebo Comparator): One drop of vehicle ophthalmic solution was instilled in both eyes TID (every six hours).
  Interventions: Other: Vehicle

INTERVENTIONS:
Drug: Oxervate — Oxervate®, an ophthalmic solution containing cenegermin 20 mcg/mL, which is a recombinant human Nerve Growth Factor (rhNGF); one drop of the test product will be instilled in both eyes three times daily (TID).
  Other Names: Cenegermin
  Arms: Oxervate
Other: Vehicle — Vehicle will be instilled with the same scheme of the test product
  Other Names: Reference product
  Arms: Vehicle

SUMMARY:
Primary objectives

* To compare the efficacy of cenegermin vs vehicle in Schirmer I test (without anaesthesia) >10mm/5min at Week 4 by testing the superiority.
* To compare the efficacy of cenegermin vs vehicle in Symptom Assessment in Dry Eye questionnaire (SANDE) global score at Week 12 by testing the superiority.

Secondary objectives

* To compare the efficacy of cenegermin vs vehicle in Schirmer I test at Week 4, 8, 12 and 16 by testing the superiority.
* To compare the efficacy of cenegermin vs vehicle in Cornea and conjunctiva vital staining with fluorescein (National Eye Institute [NEI] scales) at Week 4, 8, 12 and 16 by testing the superiority.
* To compare the efficacy of cenegermin vs vehicle in Tear Film Break-Up Time (TFBUT) at Week 4, 8, 12 and 16 by testing the superiority.
* To compare the efficacy of cenegermin vs vehicle in SANDE scores at Week 8, 12 and 16 by testing the superiority.
* To compare the efficacy of cenegermin vs vehicle in worsening in symptom scores (SANDE) and/or NEI score at Week 4 by testing the superiority.
* To compare the efficacy of cenegermin vs vehicle in impact of dry eye on everyday life (IDEEL) questionnaire at Week 4, 8, 12 and 16 by testing the superiority.

DETAILED DESCRIPTION:
This is a 4 week phase III, multicenter, double-masked, vehicle-controlled study to evaluate safety and efficacy of cenegermin ophthalmic solution at 20 mcg/mL solution versus vehicle, in patients with severe Sjogren's dry eye disease.

During the screening all procedures for inclusion and exclusion were performed. From the day of screening the patients stopped any kind of further treatment, except commercially available preservative free artificial tears provided by Sponsor.

At the end of the wash out period, patients meeting the entry criteria for this study were randomized 1:1 and treated for 4 weeks with either cenegermin ophthalmic solution 20 mcg/mL TID or vehicle TID.

During the 4 weeks of masked treatment only the administration of IMP was allowed.

During the follow up period, the patient could administer additional artificial tear eye drops, provided by Sponsor, only if strictly needed, and should document in the patient's diary the number of additional drops administered for each eye.

Patients were then followed up for efficacy and safety endpoints until week 16 and for safety endpoints until week 24.

The total duration of the study was 25 weeks including 1 week of screening.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥ 18 years
2. Patients with a confirmed diagnosis of Sjögren's syndrome or other autoimmune disease known to induce Sjögren's Dry Eye Disease (DED).
3. Patients with severe Sjögren's dry eye disease characterized by the following clinical features:

   1. Corneal and/or conjunctival staining with fluorescein using National Eye Institute (NEI) grading system ≥3
   2. SANDE questionnaire >25 mm
   3. Schirmer test I (without anaesthesia) ≥2 ≤5mm/5min
4. The same eye (eligible eye) must fulfill all the above criteria
5. Patients diagnosed with severe Sjögren's dry eye disease at least 3 months before enrolment
6. Best corrected distance visual acuity (BCDVA) score of ≥ 0.1 decimal units (20/200 Snellen value) in each eye at the time of study enrolment
7. If a female of childbearing potential, have a negative urine pregnancy test and use a highly effective method to avoid pregnancy for the duration of the trial and 30 days after the study treatment period. Males of reproductive potential should use effective contraception during treatment and 30 days after the study treatment period.
8. Only patients who satisfy all Informed Consent requirements may be included in the study. The patient and/or his/her legal representative must read, sign and date the Informed Consent document before any study-related procedures are performed. The Informed Consent Form signed by patients and/or legal representative must have been approved by the IRB/IEC for the current study
9. Patients must have the ability and willingness to comply with study procedures.

Exclusion Criteria:

1. Inability to speak and understand the local language sufficiently to understand the nature of the study, to provide written informed consent, and to allow the completion of all study assessments
2. Evidence of an active ocular infection, in either eye
3. Presence of any other ocular disorder or condition requiring topical medication during the entire duration of study in either eye
4. History of severe systemic allergy or of ocular allergy (including seasonal conjunctivitis) or chronic conjunctivitis and/or keratitis other than dry eye
5. Intraocular inflammation defined as Tyndall score >0
6. History of malignancy in the last 5 years
7. Systemic disease not stabilized within 1 month before Screening Visit (e.g. diabetes with glycemia out of range, thyroid malfunction) or judged by the investigator to be incompatible with the study (e.g. current systemic infections) or with a condition incompatible with the frequent assessment required by the study
8. Patient had a serious adverse reaction or significant hypersensitivity to any drug or chemically related compounds or had a clinically significant allergy to drugs, foods, amide local anesthetics or other materials including commercial artificial tears (in the opinion of the investigator).
9. Females of childbearing potential (those who are not surgically sterilized or post-menopausal for at least 1 year) are excluded from participation in the study if they meet any one of the following conditions:

   1. are currently pregnant or,
   2. have a positive result at the urine pregnancy test (Baseline/Day 1) or,
   3. intend to become pregnant during the study treatment period or,
   4. are breast-feeding or,
   5. are not willing to use highly effective birth control measures

   During the entire course of and 30 days after the study treatment periods
10. Any concurrent medical condition, that in the judgment of the PI, might interfere with the conduct of the study, confound the interpretation of the study results, or endanger the patient's well-being
11. Use of topical cyclosporine, or topical ophthalmic treatments of the same class, within 14 days of screening visit (day -8)
12. Use of topical corticosteroids, lifitegrast, autologous serum tears in either eye during the study (previous use not an exclusion criteria but must be discontinued at the screening visit)
13. Contact lenses, True Tear device, moisture goggles, sutureless amniotic membrane or punctum plug use during the study (previous use not an exclusion criteria but must be discontinued at the screening visit)
14. History of drug addiction or alcohol abuse in the last 2 years
15. Any prior ocular surgery (including refractive, palpebral and cataract surgery) if within 90 days before the screening visit
16. Participation in a clinical trial with a new active substance during the past 3 months
17. Participation in another clinical trial study at the same time as the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2022-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Mantelli, MD, Study Director — Dompé Farmaceutici
Locations (10):
- United States (7):
  - Lugene Eye Institute - Glendale Office, Glendale, California
  - David Wirta, M.D. & Associates, Newport Beach, California
  - The Johns Hopkins University, Baltimore, Maryland
  - Tufts University School of Medicine (TUSM) - New England Eye Center/Tufts Medical Center - Boston, Boston, Massachusetts
  - Houston Eye Associates HEA - Gramercy Location, Houston, Tennessee
  - Toyos Clinic - Nashville, Nashville, Tennessee
  - Virginia Eye Consultants (VEC) - Norfolk Office, Norfolk, Virginia
- Italy (3):
  - AOU Gaspare Rodolico - Ospedale San Marco, Catania
  - Università degli Studi di Milano - Ospedale San Giuseppe - UO Oculistica, Milan
  - AOU Policlinico Umberto I - Dipartimento Organi di Senso - Clinica Oculistica, Roma

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 126 patients ≥ 18 years with severe Sjögren's DE were assessed for eligibility. The enrolled patients (n=104) were randomized 1:1 in the study as follows: 52 patients to cenegermin and 52 to vehicle. A total of 5 patients discontinued the study prematurely: 2 patients from cenegermin group and 3 from vehicle. Regarding treatment discontinuation, a total of 5 patients discontinued the treatment prematurely: 3 patients from cenegermin and 2 from vehicle.
Period: Overall Study
Arm/Group | Oxervate | Vehicle
Started | 52 | 52
Randomized But Not Treated | 0 | 1
Safety Population (SAF) | 52 | 51
Full Analysis Set Population (FAS) | 52 | 51
Per Protocol Population (PP) | 46 | 47
Prematurely Study Discontinued | 2 | 3
Completed (study completed) | 50 | 49
Not Completed | 2 | 3
Not completed — Withdrawal of consent | 1 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Documented disease progression | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) population included all patients who were randomized and received at least one dose of the investigational product.
Groups:
- Oxervate (FAS): One drop of cenegermin 20 mcg/mL (rhNGF 20 mcg/mL) in the pharmaceutical form of ophthalmic sterile solution was instilled in both eyes three times daily (TID), every six hours.
  Oxervate: Oxervate®, an ophthalmic solution containing cenegermin 20 mcg/mL, which is a recombinant human Nerve Growth Factor (rhNGF); one drop of the test product will be instilled in both eyes three times daily (TID).
- Vehicle (FAS): One drop of vehicle ophthalmic solution was instilled in both eyes TID (every six hours).
  Vehicle: Vehicle will be instilled with the same scheme of the test product
- Total: Total of all reporting groups
Arm/Group | Oxervate (FAS) | Vehicle (FAS) | Total
Number analyzed (Participants) | 52 | 51 | 103
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 34 | 73
  >=65 years | 13 | 17 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (13.47) | 58.7 (14.10) | 57.0 (13.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 47 | 97
  Male | 2 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 43 | 39 | 82
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 8 | 7 | 15
Region of Enrollment [Number; unit: participants]
  United States | 25 | 28 | 53
  Italy | 27 | 23 | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Reaching a Value of Schirmer I Test (Without Anaesthesia) >10mm/5min at Week 4
Description: The Schirmer test type I (without anaesthesia) was performed to measure aqueous tear secretion. The rounded bend end of a sterile strip was inserted into the lower conjunctival sac over the temporal one-third of the lower eyelid margin. After 5 minutes had elapsed, the Schirmer's test strip was removed and the length of the tear absorption on the strip was measured (millimeters/5 minutes). The longer the wetted length, the healthier the status of the eye.
Time Frame: at week 4
Population: The Full Analysis Set (FAS) population consisted of all patients who were randomized and received at least one dose of the investigational product. The number of participants effectively analyzed was 51 in Cenegermin group and 50 in the Vehicle group. In fact 1 patient in Cenegermin group and 1 patient in vehicle group had imputed values of missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oxervate (FAS) | Vehicle (FAS)
Number analyzed (Participants) | 52 | 51
Participants | 19 | 2
Statistical Analysis 1: Comparison: Oxervate (FAS) vs Vehicle (FAS); It was analyzed by means of a logistic regression model adjusting by pre-defined baseline factors (treatment, gender, age class, baseline Schirmer I test value as fixed effects and site as random effect). For the imputation of missing data at week 4, a Multiple Imputation approach is adopted by performing a regression model with the baseline Schirmer I test value, gender, age class, and Schirmer I test at week 2 as explanatory variables and generating 200 datasets; Test type: Superiority — The following null hypothesis is defined on this endpoint: the number of patients reaching a value of Schirmer I test (without anaesthesia) >10mm/5min at week 4 in cenegermin (rhNGF) is lower or equal than control. The null hypothesis is rejected if the associated primary analysis p-value is lower than 0.025; p < 0.001, Regression, Logistic — P-value of treatment variable from logistic regression model on the number of patients reaching a value of Schirmer I test (without anaesthesia) >10mm/5min; Odds Ratio (OR) = 16.946, 95% CI 2-sided [3.412 to 84.165]

2. Primary Outcome: Change From Baseline in Symptoms Questionnaire (SANDE) Global Score at Week 12
Description: The SANDE questionnaire is comprised of two questions: 1) How often do your eyes feel dry and/or irritated? And 2) How severe you feel your symptoms of dryness and/or irritation are? The SANDE questionnaire uses a 100 mm horizontal line for each question to assess the extent of patients' symptoms. In this questionnaire, frequency of symptoms ranges from "rarely" (0) to "all of the time" (100) and the severity of symptoms ranges from "very mild" (0) to "very severe" (100). At each visit, patients were asked to place a mark on the two given lines based on the extent of their symptoms. The locations of the marks made by the patients on the 100 mm horizontal lines were measured in mm from left to right. The global SANDE score is calculated by multiplying the frequency score by the severity score and obtaining the square root.
  Both for total score and for frequency or severity scores, 0 is the best condition, 100 the worst condition.
  Please note that adjusted means are reported.
Time Frame: at week 12
Population: The Full Analysis Set (FAS) population consisted of all patients who were randomized and received at least one dose of the investigational product.
  Please note that adjusted means are reported.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Oxervate (FAS) | Vehicle (FAS)
Number analyzed (Participants) | 52 | 51
score on a scale | -29.5 [-42.126 to -16.930] | -25 [-37.009 to -12.926]
Statistical Analysis 1: Comparison: Oxervate (FAS) vs Vehicle (FAS); This endpoint was analyzed by means of an Analysis of Covariance with change from baseline in global SANDE Score at Week 12 as dependent variable, treatment, gender, age class, baseline global SANDE score as fixed effects and site as random effect. For missing data, Multiple Imputation approach is adopted by performing a regression model with the baseline global SANDE score, gender, age class, and intermediate global SANDE scores up to week 12 as explanatory variables and generating 200 datasets; Test type: Superiority — The following null hypothesis is defined on this endpoint: the change from baseline (reduction) in the global SANDE score at week 12 in cenegermin is lower or equal than control. The null hypothesis is rejected if the associated primary analysis p-value is lower than 0.025; p = 0.322, ANCOVA — P-value of adjusted means difference between treatments from the ANCOVA model on change from baseline in the global SANDE score; adjusted mean difference = -4.561, 95% CI 2-sided [-13.581 to 4.459]

3. Secondary Outcome: Key Secondary Outcome: Number of Patients Reaching a Value of Schirmer I Test (Without Anaesthesia) > 10mm/5min at Week 8
Description: The Schirmer test type I (without anaesthesia) was performed to measure aqueous tear secretion. The rounded bend end of a sterile strip was inserted into the lower conjunctival sac over the temporal one-third of the lower eyelid margin. After 5 minutes had elapsed, the Schirmer's test strip was removed and the length of the tear absorption on the strip was measured (millimeters/5 minutes). The longer and the wetted length, the healthier the status of the eye.
Time Frame: at Week 8
Population: The Full Analysis Set (FAS) population consisted of all patients who were randomized and received at least one dose of the investigational product. The number of participants with no imputed values for Schirmer I test at Week 8 was 49 in the IMP group and 49 in the vehicle group.
Measure: Count of Participants; unit: Participants
Arm/Group | Oxervate (FAS) | Vehicle (FAS)
Number analyzed (Participants) | 52 | 51
Participants | 18 | 2
Statistical Analysis 1: Comparison: Oxervate (FAS) vs Vehicle (FAS); This key secondary endpoint was analyzed by means of a logistic regression model with the number of patients reaching a value of Schirmer I test >10mm/5min at Week 8 as dependent variable, treatment, gender, age class and baseline Schirmer I test value as fixed effects and site as random effect; Test type: Superiority — Analysis was based on a logistic regression with the number of patients reaching a value of Schirmer I test >10mm/5min at week 8 as dependent variable, treatment, gender, age class and baseline Schirmer I test value as qualitative independent variables. Site was considered as random effects that vary randomly among patients; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 15.950, 95% CI 2-sided [3.091 to 82.310]

4. Secondary Outcome: Key Secondary Outcome: Change From Baseline in Symptoms Assessment in Dry Eye (SANDE) Score for Frequency at Week 12
Description: The SANDE questionnaire is comprised of two questions: 1) How often do your eyes feel dry and/or irritated? And 2) How severe you feel your symptoms of dryness and/or irritation are? This questionnaire uses a 100 mm horizontal line for each question to assess ocular discomfort and/or dryness experienced by the patients. In the SANDE questionnaire, frequency of symptoms ranges from "rarely" (0) to "all of the time" (100) and the severity of symptoms ranges from "very mild" (0) to "very severe" (100). At each visit, patients were asked to place a mark on the two given lines based on the extent of their symptoms. The locations of the marks made by the patients on the 100 mm horizontal lines were measured in mm from left to right and recorded. 0 was the best condition and 100 marked the worst condition. Global score from the SANDE questionnaire was calculated by multiplying the frequency score by the severity score and obtaining the square root.
  Means are adjusted means.
Time Frame: At week 12
Population: The Full Analysis Set (FAS) population consisted of all patients who were randomized and received at least one dose of the investigational product. The number of participants effectively analyzed was 49 in Cenegermin group and 49 in the Vehicle group. In fact 3 patients in Cenegermin group and 2 patients in vehicle group had imputed values of missing data via a MI approach.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Oxervate (FAS) | Vehicle (FAS)
Number analyzed (Participants) | 52 | 51
score on a scale | -24.546 [-38.261 to -10.831] | -21.793 [-34.944 to -8.643]
Statistical Analysis 1: Comparison: Oxervate (FAS) vs Vehicle (FAS); This endpoint was analyzed by means of an ANCOVA adjusting by pre-defined baseline factors (treatment, gender, age class, baseline SANDE score for severity as fixed effects and site as random effect); Test type: Superiority; p = 0.572, ANCOVA regression model — P-value of adjusted means difference between treatments from the ANCOVA model on change from baseline in SANDE score for frequency at Week 12; adjusted mean difference = -2.753, 95% CI 2-sided [-12.303 to 6.798]

5. Secondary Outcome: Key Secondary Outcome: Change From Baseline in Symptoms Assessment in Dry Eye (SANDE) Score for Severity at Week 12
Description: as for outcome 4
Time Frame: at Week 12
Population: The Full Analysis Set (FAS) population consisted of all patients who were randomized and received at least one dose of the investigational product. The number of participants effectively analyzed was 49 in Cenegermin group and 49 in the Vehicle group at Week 8 and Week 12, and 50 in Cenegermin group and 49 in Vehicle group at Week 16.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Oxervate (FAS) | Vehicle (FAS)
Number analyzed (Participants) | 52 | 51
score on a scale | -31.445 [-43.795 to -19.095] | -26.713 [-38.538 to -14.887]
Statistical Analysis 1: Comparison: Oxervate (FAS) vs Vehicle (FAS); [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.307, ANCOVA regression model — P-value of adjusted means difference between treatments from the ANCOVA model on change from baseline in SANDE score for severity at Week 12; adjusted mean difference = -4.732, 95% CI 2-sided [-13.819 to 4.354]

6. Secondary Outcome: Key Secondary Outcome: Change From Baseline in Quality of Life Module Measured by "Impact of Dry Eye on Everyday Life [IDEEL]" Questionnaire at Week 12 and at Week 4
Description: IDEEL is a 57-item questionnaire that assesses the impact of dry eye symptoms on everyday life. It is composed of 3 modules (Dry eye Quality of Life, Dry eye Treatment satisfaction & Bother, Dry eye Symptom Bother).
  This outcome is about the first module:
  Quality of Life module (27 items) is composed by 3 dimensions:
  Dimension 1 - Impact on Daily Activities, calculated by mean of the non-missing item scores 1-6 multiplied by 20. (range 0-100) Dim. 2 - Emotional Impact: calculated by mean of the non-missing item scores 10-20 multiplied by 25. (range 0-100) Dim. 3 - Impact on Work: calculated by mean of the non-missing item scores 23-27 multiplied by 25. (range 0-100) Scores for each dimension of this module ranged from 0 to 100, where higher scores indicated less impact on daily activities, on work and on emotions. No combination of dimensions scores is done.
Time Frame: At Weeks 12 and 4
Population: The Full Analysis Set (FAS) population consisted of all patients randomized, who received at least one dose of IP. 3 patients in Cenegermin group and 2 patients in vehicle group had imputed values of missing data for Impact on Daily Activities and Emotional Impact due to dry eye. For Impact on work due to dry eye the number of participants considered in the model was 30 in Cenegermin group and 34 in the Vehicle group, of which 4 and 6 had imputed values.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Oxervate (FAS) | Vehicle (FAS)
Number analyzed (Participants) | 52 | 51
score on a scale
  Impact on daily activities - week 12 | 13.301 [6.267 to 20.335] | 9.223 [2.437 to 16.008]
  Emotional impact due to dry eye - week 12 | 16.069 [7.476 to 24.661] | 10.519 [2.185 to 18.853]
  Impact on work due to dry eye - week 12: number analyzed (Participants) | 30 | 34
  Impact on work due to dry eye - week 12 | 18.619 [9.309 to 27.928] | 15.144 [6.371 to 23.916]
  Impact on daily activities - week 4 | 11.524 [5.207 to 17.842] | 9.364 [3.354 to 15.374]
  Emotional impact due to dry eye - week 4 | 14.385 [6.840 to 21.930] | 11.955 [4.732 to 19.177]
  Impact on work due to dry eye - week 4: number analyzed (Participants) | 30 | 34
  Impact on work due to dry eye - week 4 | 17.591 [8.213 to 26.969] | 14.291 [5.787 to 22.795]
Statistical Analysis 1: Comparison: Oxervate (FAS) vs Vehicle (FAS); Impact on daily activities at week 4; Test type: Superiority — Changes from baseline in each IDEEL modules scale score was analyzed using a mixed model for repeated measures (MMRM) adjusting by gender, age class, IDEEL module baseline value, treatment, visit and treatment by visit interaction. Subject was considered as a random effect. The covariance matrix used was "unstructured". Comparisons vs vehicle TID was provided using least square means at each visit and overall; p = 0.468, MMRM — P-value of Least Square (LS) means difference between treatments from the MMRM on change from baseline in IDEEL Quality of Life Module (Daily Activities) at Week 4; least square mean difference = 2.160, 95% CI 2-sided [-3.668 to 7.988]
Statistical Analysis 2: Comparison: Oxervate (FAS) vs Vehicle (FAS); Emotional Impact due to Dry eye at week 4; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.492, MMRM — P-value of LS means difference between treatments from the MMRM on change from baseline in IDEEL Quality of Life Module (Emotional Impact) at Week 4; least square mean difference = 2.431, 95% CI 2-sided [-4.500 to 9.362]
Statistical Analysis 3: Comparison: Oxervate (FAS) vs Vehicle (FAS); Impact on Work due to Dry Eye at week 4; Test type: Superiority — Changes from baseline in each IDEEL modules scale score was analyzed using a mixed model for repeated measures (MMRM). Analyses included the fixed, categorical effects of treatment, visit and treatment by visit interaction. Subject was considered as a random effect. The covariance matrix used was "unstructured". Comparisons vs vehicle TID was provided using least square means at each visit and overall. Missing data will be imputed according to the questionnaire manuals; p = 0.510, MMRM — P-value of LS means difference between treatments from the MMRM on change from baseline in IDEEL Quality of Life Module (Impact on Work) at Week 4; LS means difference = 3.300, 95% CI 2-sided [-6.511 to 13.111]
Statistical Analysis 4: Comparison: Oxervate (FAS) vs Vehicle (FAS); Quality of life - Impact on daily activities - Week 12; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.268, MMRM — P-value of LS means difference between treatments from the MMRM on change from baseline in IDEEL Quality of Life Module (Daily Activities) at Week 12; Least square mean difference = 4.078, 95% CI 2-sided [-3.142 to 11.299]
Statistical Analysis 5: Comparison: Oxervate (FAS) vs Vehicle (FAS); Quality of life - Emotional Impact due to Dry eye - Week 12; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.227, MMRM — P-value of LS means difference between treatments from the MMRM on change from baseline in IDEEL Quality of Life Module (Emotional Impact) at Week 12; least square mean difference = 5.550, 95% CI 2-sided [-3.462 to 14.562]
Statistical Analysis 6: Comparison: Oxervate (FAS) vs Vehicle (FAS); Quality of life - Impact on Work due to Dry Eye - Week 12; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.501, MMRM — P-value of LS means difference between treatments from the MMRM on change from baseline in IDEEL Quality of Life Module (Impact on Work) at Week 12; least square mean difference = 3.475, 95% CI 2-sided [-6.651 to 13.601]

7. Secondary Outcome: Key Secondary Outcome: Change From Baseline in "Treatment Satisfaction & Bother" Module Measured by "Impact of Dry Eye on Everyday Life [IDEEL]" Questionnaire at Weeks 12 and 4
Description: IDEEL is a 57-item questionnaire that assesses the impact of dry eye symptoms on everyday life. It is composed of 3 modules (Quality of Life, Treatment satisfaction & Bother, Symptom Bother).
  This outcome is about the second module:
  Treatment Satisfaction & Bother (8 items). This is composed by 2 dimensions:
  "Dim. 1" - Satisfaction with Treatment Effectiveness, calculated by mean of the non-missing item scores 2-5 multiplied by 25. (range 0-100) Dim. 2 - Treatment-Related Bother / Inconvenience calculated as the mean of the non-missing item scores 6, 8-10 multiplied by 25. (range 0-100)
  Scores for each dimension of this module range from 0 to 100, where higher scores indicate a greater satisfaction in treatment effectiveness and less treatment-related bother. No combination of dimension scores is done.
Time Frame: at Weeks 12 and 4
Population: The Full Analysis Set (FAS) population consisted of all patients who were randomized and received at least one dose of the investigational product. 3 patients in Cenegermin group and 4 patients in vehicle group had imputed values of missing data for Satisfaction with Treatment Effectiveness. For Treatment- Related Bother / Inconvenience, 4 patients in Cenegermin group and 3 patients in vehicle group had imputed values of missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Oxervate (FAS) | Vehicle (FAS)
Number analyzed (Participants) | 52 | 51
score on a scale
  Satisfaction with Treatment Effectiveness - week 12 | 12.733 [1.180 to 24.285] | 16.938 [5.033 to 28.844]
  Treatment- Related Bother / Inconvenience - week 12 | 6.482 [-0.877 to 13.842] | 4.239 [-2.942 to 11.420]
  Satisfaction with Treatment Effectiveness - week 4 | 13.879 [2.071 to 25.686] | 14.428 [3.246 to 25.609]
  Treatment- Related Bother / Inconvenience - week 4 | 9.505 [2.772 to 16.237] | 8.432 [1.840 to 15.025]
Statistical Analysis 1: Comparison: Oxervate (FAS) vs Vehicle (FAS); IDEEL Treatment satisfaction & Bother Module Satisfaction with Treatment Effectiveness - week 4; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.924, MMRM — P-value of LS means difference between treatments from the MMRM on change from baseline in IDEEL Treatment Satisfaction & Bother module (Satisfaction with Treatment Effectiveness) at Week 4; least square mean difference = -0.549, 95% CI 2-sided [-11.820 to 10.723]
Statistical Analysis 2: Comparison: Oxervate (FAS) vs Vehicle (FAS); IDEEL Treatment satisfaction & Bother Module - Treatment- Related Bother / Inconvenience - week 4; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.745, MMRM — P-value of LS means difference between treatments from the MMRM on change from baseline in IDEEL Treatment Satisfaction & Bother module (Treatment- Related Bother / Inconvenience) at Week 4; least square mean difference = 1.072, 95% CI 2-sided [-5.398 to 7.542]
Statistical Analysis 3: Comparison: Oxervate (FAS) vs Vehicle (FAS); IDEEL Treatment satisfaction & Bother Module - Satisfaction with Treatment Effectiveness - week 12; Test type: Superiority — Changes from baseline in each IDEEL modules scale score was analyzed using a mixed model for repeated measures (MMRM)adjusting by gender, age class, IDEEL module baseline value, treatment, visit and treatment by visit interaction. Subject was considered as a random effect. The covariance matrix used was "unstructured". Comparisons vs vehicle TID was provided using least square means at each visit and overall; p = 0.467, MMRM — P-value of LS means difference between treatments from the MMRM on change from baseline in IDEEL Treatment Satisfaction & Bother module (Satisfaction with Treatment Effectiveness) at Week 12; least square mean difference = -4.206, 95% CI 2-sided [-15.530 to 7.118]
Statistical Analysis 4: Comparison: Oxervate (FAS) vs Vehicle (FAS); IDEEL Treatment satisfaction & Bother Module - Treatment- Related Bother / Inconvenience - week 12; Test type: Superiority — [test comment as in outcome 7, analysis 3]; p = 0.564, MMRM — P-value of LS means difference between treatments from the MMRM on change from baseline in IDEEL Treatment Satisfaction & Bother module (Treatment- Related Bother / Inconvenience) at Week 12; least square mean difference = 2.244, 95% CI 2-sided [-5.387 to 9.874]

8. Secondary Outcome: Key Secondary Outcome: Change From Baseline in "Symptom Bother Module" Measured by "Impact of Dry Eye on Everyday Life [IDEEL]" Questionnaire at Weeks 12 and 4
Description: IDEEL is a 57-item questionnaire that assesses the impact of dry eye symptoms on everyday life. It is composed of 3 modules (Quality of Life, Treatment Satisfaction & Bother, Symptom Bother). This outcome is about the third module: Symptom Bother (20 items).
  This is composed by 1 dimension: Dry Eye Symptom-Bother (range 0-100) The Symptom Bother score is calculated if at least 50% (10 items) of the 20 items within the dimension are completed, and non-missing; otherwise the score is set to missing. The Symptom Bother score is calculated as the mean of the non-missing item scores 1-20 multiplied by 25. The higher the score the greater the symptom bother.
Time Frame: at Weeks 12 and 4
Population: The Full Analysis Set (FAS) population consisted of all patients who were randomized and received at least one dose of the investigational product. 3 patients in Cenegermin group and 2 patients in vehicle group had imputed values of missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Oxervate (FAS) | Vehicle (FAS)
Number analyzed (Participants) | 52 | 51
score on a scale
  week 12 | -16.323 [-23.582 to -9.064] | -7.533 [-14.574 to -0.493]
  week 4 | -10.241 [-16.924 to -3.557] | -9.435 [-15.876 to -2.995]
Statistical Analysis 1: Comparison: Oxervate (FAS) vs Vehicle (FAS); IDEEL - Symptom Bother module - week 4; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.802, MMRM — P-value of LS means difference between treatments from the MMRM on change from baseline in IDEEL Symptom Bother Module at Week 4; least square mean difference = -0.805, 95% CI 2-sided [-7.086 to 5.476]
Statistical Analysis 2: Comparison: Oxervate (FAS) vs Vehicle (FAS); IDEEL - Symptom Bother module - week 12; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.019, MMRM — P-value of LS means difference between treatments from the MMRM on change from baseline in IDEEL Symptom Bother Module at Week 12; least square mean difference = -8.789, 95% CI 2-sided [-16.160 to -1.418]

9. Secondary Outcome: Key Secondary Outcome: Change From Baseline in Cornea and Conjunctiva Vital Staining With Fluorescein (National Eye Institute [NEI] Scales) at Weeks 4, 8, 12
Description: The examiner compared the overall appearance of the patient's corneal staining with a reference figure, simulating the pattern of staining encountered in dry eye disease. non attempt was made to count the dots or to assess the position or confluence of the dots. The examiner selected the appropriate grade that best represented the state of corneal staining intuitionally. The grading system recommended by NEI divides the cornea into five zones (central, superior, temporal, nasal, and inferior) and for each zone, the severity of the corneal staining is graded on a scale from 0 to 3 based on a reference figure. Therefore the maximum score (worst outcome) was 15, and the minimum (best outcome) was 0.
Time Frame: At weeks 4, 8, 12
Population: The Full Analysis Set (FAS) population consisted of all patients who were randomized and received at least one dose of the investigational product. 3 patients in Cenegermin group and 2 patients in vehicle group had imputed values of missing data via a multiple imputation approach.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Oxervate (FAS) | Vehicle (FAS)
Number analyzed (Participants) | 52 | 51
score on a scale
  Week 4: number analyzed (Participants) | 51 | 50
  Week 4 | -4.107 [-5.723 to -2.490] | -2.588 [-4.118 to -1.059]
  Week 8: number analyzed (Participants) | 49 | 49
  Week 8 | -4.442 [-6.145 to -2.739] | -2.668 [-4.298 to -1.038]
  Week 12: number analyzed (Participants) | 49 | 49
  Week 12 | -3.714 [-5.522 to -1.905] | -2.490 [-4.222 to -0.758]
Statistical Analysis 1: Comparison: Oxervate (FAS) vs Vehicle (FAS); Herein Week 4 was considered. The change from baseline in Cornea and conjunctiva vital staining with fluorescein NEI scale was analyzed by means of an MMRM adjusting by pre-defined factors (gender, age class, NEI scale baseline value, treatment, visit, and treatment by visit interaction; subject was considered as a random effect); Test type: Superiority; p = 0.045, MMRM — P-value of LS means difference between treatments from the MMRM on change from baseline in Cornea and conjunctiva vital staining with fluorescein NEI scale at Week 4; least square mean difference = -1.518, 95% CI 2-sided [-3.005 to -0.031]
Statistical Analysis 2: Comparison: Oxervate (FAS) vs Vehicle (FAS); Herein Week 8 was considered. The change from baseline in Cornea and conjunctiva vital staining with fluorescein NEI scale was analyzed by means of an MMRM adjusting by pre-defined factors (gender, age class, NEI scale baseline value, treatment, visit, and treatment by visit interaction; subject was considered as a random effect); Test type: Superiority; p = 0.038, MMRM — P-value of LS means difference between treatments from the MMRM on change from baseline in Cornea and conjunctiva vital staining with fluorescein NEI scale at Week 8; least square mean difference = -1.773, 95% CI 2-sided [-3.446 to -0.101]
Statistical Analysis 3: Comparison: Oxervate (FAS) vs Vehicle (FAS); Herein Week 12 was considered. The change from baseline in Cornea and conjunctiva vital staining with fluorescein NEI scale was analyzed by means of an MMRM adjusting by pre-defined factors (gender, age class, NEI scale baseline value, treatment, visit, and treatment by visit interaction; subject was considered as a random effect); Test type: Superiority; p = 0.200, MMRM — P-value of LS means difference between treatments from the MMRM on change from baseline in Cornea and conjunctiva vital staining with fluorescein NEI scale at Week 12; least square mean difference = -1.224, 95% CI 2-sided [-3.096 to 0.649]

10. Secondary Outcome: Key Secondary Outcome: Change From Baseline in Tear Film Break-Up Time (TFBUT) at Week 4, Week 8, Week 12
Description: TFBUT was measured by determining the time to tear break-up.The TFBUT test was performed after instillation of 5 μl of 2% preservative free sodium fluorescein solution into the lower conjunctival sac of each eye. This measurement was performed within 10 seconds maximum. The TFBUT was measured twice during the first minute of instillation of the fluorescein. If the 2 readings differed by more than 2 sec., a third reading was taken. The TFBUT value was the average of the 2 or 3 measurements. Generally, a TFBUT value of 10-35 sec was considered normal. A value of less than 10 seconds may indicate tear film instability.
Time Frame: At weeks 4, 8, 12
Population: The Full Analysis Set (FAS) population consisted of all patients who were randomized and received at least one dose of the investigational product. 3 patients in Cenegermin group and 2 patients in vehicle group had imputed values of missing data using a MI approach.
Measure: Least Squares Mean (95% Confidence Interval); unit: seconds
Arm/Group | Oxervate (FAS) | Vehicle (FAS)
Number analyzed (Participants) | 52 | 51
seconds
  Week 4 | 1.808 [0.437 to 3.178] | 0.167 [-1.144 to 1.479]
  Week 8 | 2.010 [0.579 to 3.441] | 0.876 [-0.502 to 2.255]
  Week 12 | 1.973 [0.588 to 3.358] | 0.613 [-0.715 to 1.941]
Statistical Analysis 1: Comparison: Oxervate (FAS) vs Vehicle (FAS); Herein week 4 was considered. The change from baseline in TFBUT values was analyzed by means of a MMRM adjusting by pre-defined factors (gender, age class, TFBUT baseline value, treatment, visit, and treatment by visit interaction; subject was considered as a random effect); Test type: Superiority; p = 0.016, MMRM — P-value of LS means difference between treatments from the MMRM on change from baseline in TFBUT at Week 4; least square mean difference = 1.640, 95% CI 2-sided [0.300 to 2.980]
Statistical Analysis 2: Comparison: Oxervate (FAS) vs Vehicle (FAS); Herein week 8 was considered. The change from baseline in TFBUT values was analyzed by means of a MMRM adjusting by pre-defined factors (gender, age class, TFBUT baseline value, treatment, visit, and treatment by visit interaction; subject was considered as a random effect); Test type: Superiority; p = 0.129, MMRM — P-value of LS means difference between treatments from the MMRM on change from baseline in TFBUT at Week 8; least ssquare mean difference = 1.133, 95% CI 2-sided [-0.329 to 2.596]
Statistical Analysis 3: Comparison: Oxervate (FAS) vs Vehicle (FAS); Herein week 12 was considered. The change from baseline in TFBUT values was analyzed by means of a MMRM adjusting by pre-defined factors (gender, age class, TFBUT baseline value, treatment, visit, and treatment by visit interaction; subject was considered as a random effect); Test type: Superiority; p = 0.050, MMRM — P-value of LS means difference between treatments from the MMRM on change from baseline in TFBUT at Week 12; least square mean difference = 1.360, 95% CI 2-sided [-0.002 to 2.722]

11. Secondary Outcome: Change From Baseline in Schirmer I Test (Without Anaesthesia) [Time Frame: Week 4, 8, 12 and 16].
Description: The Schirmer test type I (without anaesthesia) was performed to measure aqueous tear secretion. The rounded bend end of a sterile strip was inserted into the lower conjunctival sac over the temporal one-third of the lower eyelid margin. After 5 minutes had elapsed, the Schirmer's test strip was removed and the length of the tear absorption on the strip was measured (millimeters/5 minutes). The longer, the wetted length, the healthier the status of the eye.
Time Frame: Week 4, 8, 12 and 16
Population: The Full Analysis Set (FAS) population consisted of all patients who were randomized and received at least one dose of the investigational product. The actual number of participants effectively analyzed was 51 in the IMP group and 50 in the vehicle group at Week 4, 49 in both IMP and vehicle group at Week 8 and at Week 12, and 50 in the IMP group and 49 in the vehicle group at Week 16.
Measure: Least Squares Mean (Standard Deviation); unit: millimeters
Arm/Group | Oxervate (FAS) | Vehicle (FAS)
Number analyzed (Participants) | 52 | 51
millimeters
  week 4: number analyzed (Participants) | 51 | 50
  week 4 | 5.4 (6.6) | 0.8 (2.7)
  week 8: number analyzed (Participants) | 49 | 49
  week 8 | 4.9 (6.6) | 1.4 (2.9)
  week 12: number analyzed (Participants) | 49 | 49
  week 12 | 3.8 (5.2) | 1.4 (4.1)
  week 16: number analyzed (Participants) | 50 | 49
  week 16 | 3.6 (5.1) | 1.7 (4.8)
Statistical Analysis 1: Comparison: Oxervate (FAS) vs Vehicle (FAS); Herein Week 4 was considered. Change from baseline between the two treatment groups was compared using a two-sample t-test or a Mann-Whitney-Wilcoxon (Wilson rank sum) test if normality assumption not met; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — p-value corresponds to a non-parametric Mann-Whitney-Wilcoxon (Wilcoxon rank sum) test of the comparisons between Cenegermin and Vehicle in all participants
Statistical Analysis 2: Comparison: Oxervate (FAS) vs Vehicle (FAS); Herein Week 8 was considered. Change from baseline between the two treatment groups was compared using a two-sample t-test or a Mann-Whitney-Wilcoxon (Wilson rank sum) test if normality assumption not met; Test type: Superiority; p = 0.009, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Oxervate (FAS) vs Vehicle (FAS); Herein Week 12 was considered. Change from baseline between the two treatment groups was compared using a two-sample t-test or a Mann-Whitney-Wilcoxon (Wilson rank sum) test if normality assumption not met; Test type: Superiority; p = 0.020, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 4: Comparison: Oxervate (FAS) vs Vehicle (FAS); Herein Week 16 was considered. Change from baseline between the two treatment groups was compared using a two-sample t-test or a Mann-Whitney-Wilcoxon (Wilson rank sum) test if normality assumption not met; Test type: Superiority; p = 0.022, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 11, analysis 1]

12. Secondary Outcome: Change From Baseline in Cornea and Conjunctiva Vital Staining With Fluorescein (National Eye Institute [NEI] Scales) at Week 16
Description: as for outcome 9
Time Frame: at Week 16
Population: The Full Analysis Set (FAS) population consisted of all patients who were randomized and received at least one dose of the investigational product. The number of participants effectively analyzed at weeks 8 and 12 was 49 in Cenegermin group and 49 in the Vehicle group. At week 4 the participants analyzed were 51 in Cenegermin and 50 in Vehicle group. At week 16, the number of participants analyzed were 50 in Cenegermin and 49 in Vehicle group.
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxervate (FAS) | Vehicle (FAS)
Number analyzed (Participants) | 50 | 49
score on a scale | -3.3 (4.6) | -2.7 (5.8)
Statistical Analysis 1: Comparison: Oxervate (FAS) vs Vehicle (FAS); [analysis description as in outcome 11, analysis 4]; Test type: Superiority; p = 0.065, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 11, analysis 1]

13. Secondary Outcome: Change From Baseline in Tear Film Break-Up Time (TFBUT) at Week 16
Description: as for outcome 10
Time Frame: at week 16
Population: The Full Analysis Set (FAS) population consisted of all patients who were randomized and received at least one dose of the investigational product. he number of participants effectively analyzed at weeks 8 and 12 was 49 in Cenegermin group and 49 at the Vehicle group. At week 4 the participants analyzed were 51 in Cenegermin and 50 in Vehicle group. At week 16, the number of participants analyzed were 50 in Cenegermin group and 49 in the Vehicle group.
Measure: Least Squares Mean (Standard Deviation); unit: seconds
Arm/Group | Oxervate (FAS) | Vehicle (FAS)
Number analyzed (Participants) | 50 | 49
seconds | 1.3 (3.1) | 0.4 (2.8)
Statistical Analysis 1: Comparison: Oxervate (FAS) vs Vehicle (FAS); [analysis description as in outcome 11, analysis 4]; Test type: Superiority; p = 0.125, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 11, analysis 1]

14. Secondary Outcome: Change From Baseline in Symptoms Questionnaire (SANDE) Global Score at Week 8, Week 12, Week 16
Description: The SANDE questionnaire is comprised of two questions: 1) How often do your eyes feel dry and/or irritated? And 2) How severe you feel your symptoms of dryness and/or irritation are? This questionnaire uses a 100 mm horizontal line for each question to assess ocular discomfort and/or dryness experienced by the patients. In the SANDE questionnaire, frequency of symptoms ranges from "rarely" (0) to "all of the time" (100) and the severity of symptoms ranges from "very mild" (0) to "very severe" (100). At each visit, patients were asked to place a mark on the two given lines based on the extent of their symptoms. The locations of the marks made by the patients on the 100 mm horizontal lines were measured in mm from left to right and recorded. 0 was the best condition and 100 marked the worst condition. Global score from the SANDE questionnaire was calculated by multiplying the frequency score by the severity score and obtaining the square root.
Time Frame: at Week 8, Week 12, Week 16
Population: as for outcome 5
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxervate (FAS) | Vehicle (FAS)
Number analyzed (Participants) | 52 | 51
score on a scale
  week 8: number analyzed (Participants) | 49 | 49
  week 8 | -26.0 (20.1) | -15.2 (22.1)
  week 12: number analyzed (Participants) | 49 | 49
  week 12 | -20.4 (22.0) | -15.7 (26.7)
  week 16: number analyzed (Participants) | 50 | 49
  week 16 | -15.2 (20.5) | -16.0 (25.2)
Statistical Analysis 1: Comparison: Oxervate (FAS) vs Vehicle (FAS); [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p = 0.005, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Oxervate (FAS) vs Vehicle (FAS); [analysis description as in outcome 11, analysis 3]; Test type: Superiority; p = 0.116, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Oxervate (FAS) vs Vehicle (FAS); [analysis description as in outcome 11, analysis 4]; Test type: Superiority; p = 0.864, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 11, analysis 1]

15. Secondary Outcome: Change From Baseline in Symptoms Questionnaire (SANDE) Score for Frequency at Week 8, Week 12, Week 16
Description: as for outcome 14
Time Frame: at Week 8, Week 12, Week 16
Population: as for outcome 5
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxervate (FAS) | Vehicle (FAS)
Number analyzed (Participants) | 52 | 51
score on a scale
  week 8: number analyzed (Participants) | 49 | 49
  week 8 | -27.1 (22.5) | -15.9 (24.4)
  week 12: number analyzed (Participants) | 49 | 49
  week 12 | -17.9 (23.4) | -15.7 (28.2)
  week 16: number analyzed (Participants) | 50 | 49
  week 16 | -12.5 (21.2) | -16.1 (25.6)
Statistical Analysis 1: Comparison: Oxervate (FAS) vs Vehicle (FAS); [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p = 0.011, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Oxervate (FAS) vs Vehicle (FAS); [analysis description as in outcome 11, analysis 3]; Test type: Superiority; p = 0.316, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Oxervate (FAS) vs Vehicle (FAS); [analysis description as in outcome 11, analysis 4]; Test type: Superiority; p = 0.685, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 11, analysis 1]

16. Secondary Outcome: Change From Baseline in Symptoms Assessment in Dry Eye (SANDE) Score for Severity at Week 8, Week 12 and Week 16
Description: as for outcome 14
Time Frame: at Week 8, week 12 and week 16
Population: as for outcome 5
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxervate (FAS) | Vehicle (FAS)
Number analyzed (Participants) | 52 | 51
score on a scale
  week 8: number analyzed (Participants) | 49 | 49
  week 8 | -23.7 (20.8) | -14.4 (21.6)
  week 12: number analyzed (Participants) | 49 | 49
  week 12 | -21.2 (23.5) | -15.7 (26.5)
  week 16: number analyzed (Participants) | 50 | 49
  week 16 | -16.6 (23.6) | -16.1 (25.9)
Statistical Analysis 1: Comparison: Oxervate (FAS) vs Vehicle (FAS); [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p = 0.016, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Oxervate (FAS) vs Vehicle (FAS); [analysis description as in outcome 11, analysis 3]; Test type: Superiority; p = 0.160, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Oxervate (FAS) vs Vehicle (FAS); [analysis description as in outcome 11, analysis 4]; Test type: Superiority; p = 0.839, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 11, analysis 1]

17. Secondary Outcome: Number of Patients Who Experienced a Worsening in Symptoms Scores (SANDE) and/or NEI Score > = 50% at Week 4
Description: Symptoms Scores (SANDE) and/or NEI Score were punctually described in the previous outcome descriptions.
  For Sande score, the scale ranges from 0 to 100 for both severity and frequency, where 0 was the best condition and 100 marked the worst condition. Hence the higher the score, the worse the outcome.
  For NEI score, the maximum score (worst outcome) was 15, and the minimum (best outcome) was 0; hence the higher the score, the worse the outcome.
Time Frame: at week 4
Population: The Full Analysis Set (FAS) population consisted of all patients who were randomized and received at least one dose of the investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Oxervate (FAS) | Vehicle (FAS)
Number analyzed (Participants) | 52 | 51
Participants | 4 | 11
Statistical Analysis 1: Comparison: Oxervate (FAS) vs Vehicle (FAS); Test type: Superiority; p = 0.0455, Chi-squared

18. Secondary Outcome: Change From Baseline in Quality of Life Module Measured by "Impact of Dry Eye on Everyday Life [IDEEL]" Questionnaire at Weeks 8 and 16
Description: as for outcome 6
Time Frame: At weeks 8 and 16
Population: The Full Analysis Set (FAS) consisted of all patients randomized and dosed with at least one dose of the IP. The # of pts actually analyzed for Impact on Daily Activities and Emotional Impact due to Dry Eye was:
  Week 4:
  n=51 Cenegermin (C) n=50 Vehicle (V);
  Weeks 8 and 12:
  n=49 in both groups
  Week 16:
  n=50 C n=49 V.
  For Impact on work due to dry eye the No of pts actually analyzed was:
  Weeks 4 and 8 n= 24 C n= 30 V Week 12 n=23 C n=28 V
  Week 16:
  n= 23 C n=29 V
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxervate (FAS) | Vehicle (FAS)
Number analyzed (Participants) | 52 | 51
score on a scale
  Impact on Daily Activities - week 8: number analyzed (Participants) | 49 | 49
  Impact on Daily Activities - week 8 | 14.6 (18.8) | 6.5 (23.2)
  Emotional Impact due to Dry Eye - week 8: number analyzed (Participants) | 49 | 49
  Emotional Impact due to Dry Eye - week 8 | 18.4 (21.9) | 10.3 (22.9)
  Impact on Work due to Dry Eye - week 8: number analyzed (Participants) | 24 | 30
  Impact on Work due to Dry Eye - week 8 | 17.7 (25.7) | 9.5 (25.9)
  Impact on Daily Activities - week 16: number analyzed (Participants) | 50 | 49
  Impact on Daily Activities - week 16 | 15.1 (20.8) | 9.7 (21.1)
  Emotional Impact due to Dry Eye - week 16: number analyzed (Participants) | 50 | 49
  Emotional Impact due to Dry Eye - week 16 | 19.0 (23.1) | 11.5 (23.3)
  Impact on Work due to Dry Eye - week 16: number analyzed (Participants) | 23 | 29
  Impact on Work due to Dry Eye - week 16 | 20.9 (24.2) | 9.3 (26.7)
Statistical Analysis 1: Comparison: Oxervate (FAS) vs Vehicle (FAS); Quality of life - Impact on daily activities - Week 8; Test type: Superiority — Changes from baseline in each IDEEL modules scale score was analyzed by comparing the two treatment groups using a two-sample t-test or a Mann-Whitney-Wilcoxon (Wilson rank sum) test if normality assumption was not met; p = 0.060, t-test, 2 sided — p-value corresponds to two sample (independent group) t-test of the comparisons between Cenegermin and Vehicle in all participants
Statistical Analysis 2: Comparison: Oxervate (FAS) vs Vehicle (FAS); Quality of life - Emotional impact due to Dry eye - Week 8; Test type: Superiority — [test comment as in outcome 18, analysis 1]; p = 0.079, t-test, 2 sided — [p-value comment as in outcome 18, analysis 1]
Statistical Analysis 3: Comparison: Oxervate (FAS) vs Vehicle (FAS); Quality of life - Impact on work due to Dry Eye - Week 8; Test type: Superiority — [test comment as in outcome 18, analysis 1]; p = 0.251, t-test, 2 sided — [p-value comment as in outcome 18, analysis 1]
Statistical Analysis 4: Comparison: Oxervate (FAS) vs Vehicle (FAS); Quality of life - Impact on daily activities - Week 16; Test type: Superiority — [test comment as in outcome 18, analysis 1]; p = 0.203, t-test, 2 sided — [p-value comment as in outcome 18, analysis 1]
Statistical Analysis 5: Comparison: Oxervate (FAS) vs Vehicle (FAS); Quality of life - Emotional impact due to Dry eye - Week 16; Test type: Superiority — [test comment as in outcome 18, analysis 1]; p = 0.114, t-test, 2 sided — [p-value comment as in outcome 18, analysis 1]
Statistical Analysis 6: Comparison: Oxervate (FAS) vs Vehicle (FAS); Quality of life - Impact on work due to Dry Eye - Week 16; Test type: Superiority — [test comment as in outcome 18, analysis 1]; p = 0.112, t-test, 2 sided — [p-value comment as in outcome 18, analysis 1]

19. Secondary Outcome: Change From Baseline in "Symptom Bother Module" Measured by "Impact of Dry Eye on Everyday Life [IDEEL]" Questionnaire at Week 8 and Week 16
Description: as for outcome 8
Time Frame: at Week 8 and Week 16
Population: The Full Analysis Set (FAS) population consisted of all patients who were randomized and received at least one dose of the investigational product. The number of participants effectively analyzed was 51 in Cenegermin group and 50 in the Vehicle group at Week 4, 49 in both treatment groups at Week 8 and Week 12, 50 in Cenegermin group and 49 in Vehicle group at Week 16.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxervate (FAS) | Vehicle (FAS)
Number analyzed (Participants) | 52 | 51
score on a scale
  week 8: number analyzed (Participants) | 49 | 49
  week 8 | -19.5 (20.3) | -6.9 (19.2)
  week 16: number analyzed (Participants) | 50 | 49
  week 16 | -18.6 (19.4) | -11.1 (22.3)
Statistical Analysis 1: Comparison: Oxervate (FAS) vs Vehicle (FAS); Symptom bother module - Week 8; Test type: Superiority — [test comment as in outcome 18, analysis 1]; p = 0.002, t-test, 2 sided — [p-value comment as in outcome 18, analysis 1]
Statistical Analysis 2: Comparison: Oxervate (FAS) vs Vehicle (FAS); Symptom bother module - Week 16; Test type: Superiority — [test comment as in outcome 18, analysis 1]; p = 0.076, t-test, 2 sided — [p-value comment as in outcome 18, analysis 1]

20. Secondary Outcome: Change From Baseline in "Treatment Satisfaction & Bother" Module Measured by "Impact of Dry Eye on Everyday Life [IDEEL]" Questionnaire at Week 8 and Week 16
Description: IDEEL is a 57-item questionnaire that assesses the impact of dry eye symptoms on everyday life. It is composed of 3 modules (Quality of Life, Treatment satisfaction & Bother, Symptom Bother).
  This outcome is about the second module:
  Treatment Satisfaction & Bother (8 items). This is composed by 2 dimensions:
  Dim. 1 - Satisfaction with Treatment Effectiveness, calculated by mean of the non-missing item scores 2-5 multiplied by 25. (range 0-100) Dim. 2 - Treatment-Related Bother / Inconvenience calculated as the mean of the non-missing item scores 6, 8-10 multiplied by 25. (range 0-100)
  Scores for each dimension of this module range from 0 to 100, where higher scores indicate a greater satisfaction in treatment effectiveness and less treatment-related bother. No combination of dimension scores is done.
Time Frame: at Week 8 and Week 16
Population: The FAS consisted of all patients randomized and dosed with at least one dose of the IP. The # of pts effectively analyzed for Impact on Daily Activities and Emotional Impact due to Dry Eye was:
  for Satisfaction with Treatment Effectiveness section:
  Wk 4:
  n=48 C n=44 V;
  Wk 8:
  n=47 C n=44 V Wk 12 n=48 C n=44 V
  Wk 16:
  n=48 C n=42 V.
  For T-Related Bother / Inconvenience section:
  Wk 4 n= 48 C n= 44 V
  Wk 8:
  n=46 both groups Wk 12 n=47 C n=46 V
  Wk 16:
  n= 48 C n=46 V
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxervate (FAS) | Vehicle (FAS)
Number analyzed (Participants) | 52 | 51
score on a scale
  Satisfaction with Treatment Effectiveness - week 8: number analyzed (Participants) | 47 | 44
  Satisfaction with Treatment Effectiveness - week 8 | 17.7 (31.0) | 7.7 (36.4)
  Treatment- Related Bother / Inconvenience - week 8: number analyzed (Participants) | 46 | 46
  Treatment- Related Bother / Inconvenience - week 8 | 16.6 (21.1) | 2.7 (28.1)
  Satisfaction with Treatment Effectiveness - week 16: number analyzed (Participants) | 48 | 42
  Satisfaction with Treatment Effectiveness - week 16 | 13.4 (28.7) | 1.2 (35.9)
  Treatment- Related Bother / Inconvenience - week 16: number analyzed (Participants) | 48 | 46
  Treatment- Related Bother / Inconvenience - week 16 | 13.3 (23.6) | 5.3 (27.3)
Statistical Analysis 1: Comparison: Oxervate (FAS) vs Vehicle (FAS); IDEEL - Satisfaction with Treatment Effectiveness - Week 8; Test type: Superiority — [test comment as in outcome 18, analysis 1]; p = 0.160, t-test, 2 sided — [p-value comment as in outcome 18, analysis 1]
Statistical Analysis 2: Comparison: Oxervate (FAS) vs Vehicle (FAS); IDEEL - Treatment- Related Bother / Inconvenience - Week 8; Test type: Superiority — [test comment as in outcome 18, analysis 1]; p = 0.009, t-test, 2 sided — [p-value comment as in outcome 18, analysis 1]
Statistical Analysis 3: Comparison: Oxervate (FAS) vs Vehicle (FAS); IDEEL - Satisfaction with Treatment Effectiveness - Week 16; Test type: Superiority — [test comment as in outcome 18, analysis 1]; p = 0.076, t-test, 2 sided — [p-value comment as in outcome 18, analysis 1]
Statistical Analysis 4: Comparison: Oxervate (FAS) vs Vehicle (FAS); IDEEL - Treatment- Related Bother / Inconvenience - Week 16; Test type: Superiority — [test comment as in outcome 18, analysis 1]; p = 0.128, t-test, 2 sided — [p-value comment as in outcome 18, analysis 1]

21. Other Pre Specified Outcome: Incidence and Frequency of TEAEs, Assessed Throughout the Study.
Description: TEAE=any AE started on or after the date of the first dose of study medication or started prior to first dose and worsened in severity after the first dose.
Time Frame: From Screening to Visit 7 (follow-up, week 24)
Population: The SAF population consisted of all randomized patients who received at least one dose of the investigational product. SAF set was analysed according to the actual treatment received. The SAF population was used to present results on safety data.
Measure: Count of Participants; unit: Participants
Groups:
- Oxervate (SAF): One drop of cenegermin 20 mcg/mL (rhNGF 20 mcg/mL) in the pharmaceutical form of ophthalmic sterile solution was instilled in both eyes three times daily (TID), every six hours.
  Oxervate: Oxervate®, an ophthalmic solution containing cenegermin 20 mcg/mL, which is a recombinant human Nerve Growth Factor (rhNGF); one drop of the test product will be instilled in both eyes three times daily (TID).
- Vehicle (SAF): One drop of vehicle ophthalmic solution was instilled in both eyes TID (every six hours).
  Vehicle: Vehicle will be instilled with the same scheme of the test product
Arm/Group | Oxervate (SAF) | Vehicle (SAF)
Number analyzed (Participants) | 52 | 51
Participants
  TEAE - Ophtalmic | 35 | 13
  TEAE - Non Ophtalmic | 16 | 9
  Severe TEAE - Ophtamic | 5 | 1
  Severe TEAE - Non Opthalmic | 2 | 1
  Serious TEAE - Ophtalmic | 1 | 0
  Serious TEAE - Non Ophtalmic | 2 | 1
  non-serious TEAE | 37 | 15
  Adverse Drug Reaction (ADR) - Ophtalmic | 34 | 8
  Adverse Drug Reaction - Non Ophtalmic | 4 | 2
  Serious ADR | 1 | 0
  TEAE leading to IMP discontinuation | 2 | 1
  TEAE leading to study discontinuation | 0 | 1
  TEAE leading to death | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from screening visit (Day -8) to follow up (Day 168+/- 7 days)
Description: Adverse Event (AE) was defined as any untoward medical occurrence in a patient or clinical investigation subject administered a medicinal product and which did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.
Arm/Group | Oxervate (SAF) | Vehicle (SAF)
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/51
Serious Adverse Events (participants affected / at risk) | 2/52 | 1/51
Other Adverse Events (participants affected / at risk) | 37/52 | 15/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxervate (SAF) (N=52) | Vehicle (SAF) (N=51)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxervate (SAF) (N=52) | Vehicle (SAF) (N=51)
Anaemia - Mild (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Deafness bilateral - Mild (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo positional - Moderate (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Asthenopia - Mild (Eye disorders) | 1 (1) | 1 (1)
Chalazion - Mild (Eye disorders) | 1 (1) | 0 (0)
Chalazion - Moderate (Eye disorders) | 1 (1) | 0 (0)
Conjunctival hyperaemia - Mild (Eye disorders) | 1 (1) | 0 (0)
Corneal epithelium defect - Mild (Eye disorders) | 0 (0) | 1 (1)
Corneal oedema - Moderate (Eye disorders) | 1 (1) | 0 (0)
Dry eye - Mild (Eye disorders) | 2 (2) | 0 (0)
Dry eye - Moderate (Eye disorders) | 2 (2) | 1 (2)
Erythema of eyelid - Mild (Eye disorders) | 0 (0) | 1 (1)
Eye discharge - Mild (Eye disorders) | 2 (2) | 1 (1)
Eye discharge - Moderate (Eye disorders) | 0 (0) | 1 (1)
Eye inflammation - Moderate (Eye disorders) | 0 (0) | 1 (1)
Eye irritation - Mild (Eye disorders) | 1 (2) | 1 (2)
Eye irritation - Moderate (Eye disorders) | 1 (2) | 2 (2)
Eye pain - Mild (Eye disorders) | 16 (19) | 3 (3)
Eye pain - Moderate (Eye disorders) | 7 (8) | 2 (2)
Eye pain - Severe (Eye disorders) | 3 (4) | 0 (0)
Eye pruritus - Mild (Eye disorders) | 1 (1) | 4 (5)
Eye pruritus - Moderate (Eye disorders) | 0 (0) | 2 (2)
Eyelid disorder - Mild (Eye disorders) | 1 (1) | 0 (0)
Eyelid margin crusting - Mild (Eye disorders) | 0 (0) | 1 (1)
Eyelid pain - Mild (Eye disorders) | 6 (9) | 0 (0)
Eyelid pain - Moderate (Eye disorders) | 5 (5) | 0 (0)
Eyelid pain - Severe (Eye disorders) | 1 (2) | 0 (0)
Eyelid ptosis - Moderate (Eye disorders) | 1 (1) | 0 (0)
Eyelid sensory disorder - Mild (Eye disorders) | 1 (1) | 0 (0)
Foreign body sensation in eyes - Mild (Eye disorders) | 0 (0) | 1 (1)
Foreign body sensation in eyes - Moderate (Eye disorders) | 2 (2) | 3 (3)
Keratopathy - Moderate (Eye disorders) | 1 (1) | 0 (0)
Lacrimation increased - Mild (Eye disorders) | 1 (1) | 0 (0)
Ocular hyperaemia - Mild (Eye disorders) | 1 (1) | 2 (2)
Periorbital pain - Mild (Eye disorders) | 1 (1) | 0 (0)
Periorbital pain - Moderate (Eye disorders) | 1 (1) | 0 (0)
Photophobia - Mild (Eye disorders) | 1 (1) | 1 (1)
Photophobia - Moderate (Eye disorders) | 1 (1) | 1 (1)
Photophobia - Severe (Eye disorders) | 2 (2) | 1 (1)
Punctate keratitis - Moderate (Eye disorders) | 1 (1) | 0 (0)
Swelling of eyelid - Moderate (Eye disorders) | 1 (1) | 0 (0)
Ulcerative keratitis - Mild (Eye disorders) | 1 (1) | 0 (0)
Vision blurred - Mild (Eye disorders) | 2 (2) | 1 (1)
Vision blurred - Moderate (Eye disorders) | 2 (2) | 1 (1)
Visual acuity reduced - Moderate (Eye disorders) | 1 (1) | 0 (0)
Visual field defect - Mild (Eye disorders) | 1 (1) | 0 (0)
Visual impairment - Moderate (Eye disorders) | 1 (1) | 1 (1)
Pancreatitis acute - Moderate (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue - Severe (General disorders) | 1 (1) | 0 (0)
Instillation site pain - Mild (General disorders) | 1 (1) | 0 (0)
Bile duct stone - Moderate (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypertransaminasaemia - Moderate (Hepatobiliary disorders) | 1 (1) | 0 (0)
Seasonal allergy - Moderate (Immune system disorders) | 0 (0) | 2 (2)
Bacteraemia - Moderate (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 - Mild (Infections and infestations) | 1 (1) | 1 (1)
COVID-19 - Moderate (Infections and infestations) | 1 (1) | 0 (0)
Coronavirus infection - Mild (Infections and infestations) | 0 (0) | 1 (1)
Genital herpes simplex -Mild (Infections and infestations) | 1 (2) | 0 (0)
Otitis media - Mild (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis - Mild (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection - Mild (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection - Mild (Infections and infestations) | 1 (1) | 1 (1)
Arthropod bite - Mild (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus injury - Moderate (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration - Moderate (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture - Mild (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone increased - Mild (Investigations) | 1 (1) | 0 (0)
Arthralgia - Moderate (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Arthropathy - Severe (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain - Mild (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fibromyalgia - Moderate (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in jaw - Moderate (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rheumatoid arthritis - Mild (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Scleroderma - Moderate (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sjogren's syndrome - Moderate (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Systemic lupus erythematosus - Moderate (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Aura - Mild (Nervous system disorders) | 1 (1) | 0 (0)
Headache - Mild (Nervous system disorders) | 1 (1) | 1 (1)
Headache - Moderate (Nervous system disorders) | 1 (1) | 1 (2)
Headache - Severe (Nervous system disorders) | 1 (1) | 0 (0)
Migraine - Mild (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-01-26): https://cdn.clinicaltrials.gov/large-docs/80/NCT05133180/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-14): https://cdn.clinicaltrials.gov/large-docs/80/NCT05133180/SAP_001.pdf